CLINICAL TRIAL: NCT06506721
Title: Balloon Catheter vs. Hygroscopic Cervical Dilator for Labour Induction After Previous Caesarean Section: an Open Prospective Randomized Controlled Trial
Brief Title: Comparison Between Two Medical Devices for Labor Induction After Previous C-section
Acronym: DiBal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1650; 10000993 (Other: Swissmedic); 2019-02112 (Other: Cantonal Ethics Committee of Bern); CIV-21-12-038486 (Other: EUDAMED)
Record Dates: First submitted 2024-06-24; First posted 2024-07-17 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Delivery, Obstetric; Cesarean Section; Obstetric Delivery
Keywords: Trial of Labour

STUDY DESIGN:
Intervention Model Description: Open (unblinded) prospective randomized trial
Masking Description: due to nature of the induction method, blinding of women an/ or doctors is considered non-feasible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double balloon device (Active Comparator): In this group of patients, the labour will be induced using the Cook double balloon device
  Interventions: Device: Double ballon device, Cook
- Hygroscopic cervix dilators (Active Comparator): In this group of patients, the labour will be induced using the hygroscopic cervix dilators Dilapan-S
  Interventions: Device: Hygroscopic cervix dilators, Dilapan-S

INTERVENTIONS:
Device: Double ballon device, Cook — Cook double balloon will be introduced transcervically. The double balloon will be inflated with sterile 0-9% saline solution (maximum 80 ml in each balloon of the double device), then the catheter will be fixed with a tape at the women's thigh without traction. The catheter will remain in place until spontaneously expelled or start of active labour.
  If neither happens, the device will be removed after 12-24 hours and oxytocin will be administered and amniotomy as soon as feasible. If the cervix remains unfavorable after two cycles of 6 hours of oxytocin infusion, the induction will be classified as unsuccessful and C-section will be performed.
  Arms: Double balloon device
Device: Hygroscopic cervix dilators, Dilapan-S — A maximum number of 5 hygroscopic cervical dilator rods will be inserted transcervically, after humidification with sterile 0.9% saline solution. They will be fixed in this position by inserting a humidified compress into the vagina. They will remain in place until spontaneously expelled or until start of active labour.
  In neither happens, the devices will be removed after 12-24 hours and oxytocin will be administered and amniotomy as soon as feasible. If the cervix remains unfavorable after two cycles of 6 hours of oxytocin infusion, the induction will be classified as unsuccessful and C-section will be performed.
  Arms: Hygroscopic cervix dilators

SUMMARY:
The objective of the study ist to compare the Dilapan-S and the Cook Ballon device for the mechanical induction of labour in women with a previous C-section. There is currently lack of data regarding this comparison of the two methods for mechanical labour induction in this patient collective. Any method used for labour induction is therefore off-label. The primary outcome is the time between placement of the device and delivery. Ad secondary outcomes are among others the cesarean delivery rate and patient satisfaction with the induction method.

DETAILED DESCRIPTION:
The cesarean section (CS) rate is increasing worldwide, with previous CS being an important factor contributing to this trend. The investigators think that VBAC may be safe, provided a careful selection of the patients is performed. The individual birth management is particularly important if labour has to be induced, as in case of approximately 25% of women attempting VBAC. Counselling patients about labour induction can be challenging, as they should be offered not only a safe, but also an effective method. Labor induction can be achieved by using several approaches: administration of drugs, which induce uterine contractions, such as prostaglandins or oxytocin, performing an amniotomy, or using mechanical methods. In Switzerland and implicitly in the investigators' institution, PGE after CS are rarely employed in carefully selected cases. Oxytocin administration after performing amniotomy is considered to be a safe method, but may be less effective with an unfavorable BISHOP score (<6).

An possible alternative in case of unripe cervix is induction of labour by use of mechanical methods: balloon catheters and laminaria stents. The investigators currently use the double balloon catheter device (Cook Inc) for this purpose. This device is inserted transcervically and both ballons are inflated with sterile 0.9% saline solution. The catheter remains in place until spontaneously expelled or until start of active labour. If neither happens, it will be removed after 12 hours, followed by oxytocin administration and amniotomy.

Recently, an alternative method for mechanical induction is gaining increased attention: the use of hygroscopic cervical dilators. The method seems to be equally effective and safe as directly compared to a single device catheter in a low risk population of women without uterine scar. When used in patients with previous cesarean section, the rate of spontaneous labour seems to resemble existent data for induction with balloon catheter, this including the investigators' collective.

One of the advantages of Dilapan-S® could be the lack of vaginal protrusion and the fact that it does not have to be fixated under tension. Women seem to feel more mobile with Dilapan®, the perception of relaxation moments between contractions as well as sleep periods during the induction seem to be improved with Dilapan®.

ELIGIBILITY:
Inclusion Criteria:

* All women >= 18years old with a previous CS and an indication of labour induction, between 24-42 weeks of pregnancy.
* Modified Bishop-Score < 6
* Informed consent

Exclusion criteria:

* More than 1 CS
* Premature rupture of membranes
* Vaginal infection
* Intrauterine fetal demise
* Twin pregnancy
* Contraindication against labour induction or vaginal delivery
* Vaginal bleeding
* Simultaneous external administration of prostaglandins planned
* Placenta praevia, vasa praevia or placenta accreta spectrum
* Transverse fetal orientation
* Prolapsed umbilical cord
* Prior hysterotomy, classic uterine incision, myomectomy or any other full thickness uterine incision (except C-section)
* Pelvic structural anomaly
* Active genital herpes infection
* Invasive cervical cancer
* Abnormal fetal heart rate pattern
* Breech presentation
* Maternal heart disease
* Polyhydramnios
* Presentic part above the pelvic inlet
* Severe maternal hypertension

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 137 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Induction-to-delivery interval (IDI) after induction of labour (COOK catheter or Dilapan) in women with previous CS. | 72 hours
  The time between placement of the device and delivery

SECONDARY OUTCOMES:
Cesarean delivery rate | 72 hours
  How many women will get at the end a C-section after inducing the labour
Neonatal outcomes | 2 hours
  The cord arterial pH (< 7.10)
Neonatal outcomes | 2 hours
  5 minutes APGAR-Score (< 7)
Neonatal outcomes | 2 hours
  Transfer to the ICU
Maternal infection rate | 96 hours
  To asses the maternal infection status the investigators use the temperature (fever >38.0°), Leucocytosis (> 16.000 G/l), CRP (> 50)
Patient satisfaction | 96 hours
  All participant will receive a questionnaire after birth regarding the time from induction initiation until active phase of labour, covering questions such as convenience of the induction method (multiplicity of vaginal manipulation, comfort and pain experience)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Surbek, Prof. Dr., Principal Investigator — Co-Chairman, Departament of Obstetrics an Gynäkology, Head of Obstetrics and feto-maternal Medicine, University Hospital Bern
Locations (1):
- University Hospital of Obstetrics and Gynäkologie, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists Committee on Obstetric Practice. ACOG Committee Opinion No. 342: induction of labor for vaginal birth after cesarean delivery. Obstet Gynecol. 2006 Aug;108(2):465-8. doi: 10.1097/00006250-200608000-00045. PMID 16880321
- [Background] Menacker F, Declercq E, Macdorman MF. Cesarean delivery: background, trends, and epidemiology. Semin Perinatol. 2006 Oct;30(5):235-41. doi: 10.1053/j.semperi.2006.07.002. PMID 17011392
- [Background] Greene MF. Vaginal birth after cesarean revisited. N Engl J Med. 2004 Dec 16;351(25):2647-9. doi: 10.1056/NEJMe048277. Epub 2004 Dec 14. No abstract available. PMID 15598961
- [Background] American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, Cahill AG, Guise JM, Rouse DJ. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol. 2014 Mar;210(3):179-93. doi: 10.1016/j.ajog.2014.01.026. PMID 24565430
- [Background] Martel MJ, MacKinnon CJ; Clinical Practice Obstetrics Committee, Society of Obstetricians and Gynaecologists of Canada. Guidelines for vaginal birth after previous Caesarean birth. J Obstet Gynaecol Can. 2005 Feb;27(2):164-88. doi: 10.1016/s1701-2163(16)30188-8. English, French. PMID 15943001
- [Background] Ravasia DJ, Wood SL, Pollard JK. Uterine rupture during induced trial of labor among women with previous cesarean delivery. Am J Obstet Gynecol. 2000 Nov;183(5):1176-9. doi: 10.1067/mob.2000.109037. PMID 11084562
- [Background] Grobman WA, Gilbert S, Landon MB, Spong CY, Leveno KJ, Rouse DJ, Varner MW, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, O'Sullivan MJ, Sibai BM, Langer O, Thorp JM, Ramin SM, Mercer BM. Outcomes of induction of labor after one prior cesarean. Obstet Gynecol. 2007 Feb;109(2 Pt 1):262-9. doi: 10.1097/01.AOG.0000254169.49346.e9. PMID 17267822
- [Background] Saad AF, Villarreal J, Eid J, Spencer N, Ellis V, Hankins GD, Saade GR. A randomized controlled trial of Dilapan-S vs Foley balloon for preinduction cervical ripening (DILAFOL trial). Am J Obstet Gynecol. 2019 Mar;220(3):275.e1-275.e9. doi: 10.1016/j.ajog.2019.01.008. Epub 2019 Feb 18. PMID 30790569
- [Background] Radan AP, Amylidi-Mohr S, Mosimann B, Simillion C, Raio L, Mueller M, Surbek D. Safety and effectiveness of labour induction after caesarean section using balloon catheter or oxytocin. Swiss Med Wkly. 2017 Nov 8;147:w14532. doi: 10.4414/smw.2017.14532. eCollection 2017. PMID 29120029
- [Background] Gupta J, Chodankar R, Baev O, Bahlmann F, Brega E, Gala A, Hellmeyer L, Hruban L, Maier J, Mehta P, Murthy A, Ritter M, Saad A, Shmakov R, Suneja A, Zahumensky J, Gdovinova D. Synthetic osmotic dilators in the induction of labour-An international multicentre observational study. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:70-75. doi: 10.1016/j.ejogrb.2018.08.004. Epub 2018 Aug 3. PMID 30107363
- [Background] Koenigbauer JT, Schalinski E, Jarchau U, Gauger U, Brandt K, Klaucke S, Scharf JP, Rath W, Hellmeyer L. Cervical ripening after cesarean section: a prospective dual center study comparing a mechanical osmotic dilator vs. prostaglandin E2. J Perinat Med. 2021 Aug 2;49(7):797-805. doi: 10.1515/jpm-2021-0157. Print 2021 Sep 27. PMID 34333894
- [Result] Mueller M, Kolly L, Bauman M, Imboden S, Surbek D. Analysis of caesarean section rates over time in a single Swiss centre using a ten-group classification system. Swiss Med Wkly. 2014 Feb 19;144:w13921. doi: 10.4414/smw.2014.13921. PMID 24554332
- [Result] Hamilton BE, Martin JA, Osterman MJ, Curtin SC, Matthews TJ. Births: Final Data for 2014. Natl Vital Stat Rep. 2015 Dec;64(12):1-64. PMID 26727629
- [Result] Christmann-Schmid C, Raio L, Scheibner K, Muller M, Surbek D. Back to "once a caesarean: always a caesarean"? A trend analysis in Switzerland. Arch Gynecol Obstet. 2016 Nov;294(5):905-910. doi: 10.1007/s00404-016-4055-4. Epub 2016 Mar 15. PMID 26980229
- See also: Surbek D, Rath W. Vaginale Geburt nach vorausgegangener Sectio - riskant? — https://www.thieme-connect.de/products/ejournals/abstract/10.1055/s-2006-924757
- See also: Geburtseinleitung bei Zustand nach Sectio — https://www.thieme-connect.de/products/ejournals/abstract/10.1055/s-2006-924756
- See also: Dilapan Information for patients — https://www.dilapan.com/